CLINICAL TRIAL: NCT00686517
Title: An Open, Randomized, Multicentre Trial to Evaluate Efficacy and Safety of a 24-week Course of PEG-Interferon Alpha-2b Versus a 12-week Course of PEG-Interferon Alpha-2b Alone or Plus Ribavirin in Patients With Acute Hepatitis C
Brief Title: Evaluation of Peginterferon Alfa-2b Monotherapy and Combination With Ribavirin in Participants With Acute Hepatitis C (P03552/MK-4031-137)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Bioikos Ambiente Srl (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03552
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2012-01-31 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG-IFN 24 (Experimental): pegylated interferon alpha-2b 1.5 ug/kg/week for 24 weeks
  Interventions: Biological: Pegylated interferon alfa-2b
- PEG-IFN 12 (Experimental): pegylated interferon alpha-2b 1.5 ug/kg/week for 12 weeks
  Interventions: Biological: Pegylated interferon alfa-2b
- PEG-IFN + RVB 12 (Experimental): pegylated interferon alpha-2b 1.5 ug/kg/week in combination with ribavirin at the dose of 10.6 mg/kg/day for 12 weeks
  Interventions: Biological: Pegylated interferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Biological: Pegylated interferon alfa-2b — 1.5 ug/kg/week SC for 12 or 24 weeks
  Other Names: SCH 54031, PegIntron
Drug: Ribavirin — Ribavirin at the dose of 10.6 mg/kg/day for 12 weeks
  Other Names: SCH 18908, Rebetol
  Arms: PEG-IFN + RVB 12

SUMMARY:
The objective of this study is to evaluate the efficacy of three regimens of pegylated interferon-alfa 2b (PEG-IFN) either as monotherapy or in combination with ribavirin in participants with acute hepatitis C. After 12 weeks of observation from disease onset, participants will receive one of the following regimens: (1) a 24-week course of PEG-IFN monotherapy (PEG-IFN 24); or (2) a 12-week course of PEG-IFN monotherapy (PEG-IFN-12); or (3) a 12-week course of PEG-IFN in combination with ribavirin (PEG-IFN + RVB 12). After the treatment period, participants will enter a 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute hepatitis C virus (HCV).
* Normal and Elevated serum alanine transferase (ALT) levels
* Positive serum HCV-RNA.
* Aged between 18 and 65 years.
* Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of the drug. Additionally, all fertile males with partners of childbearing age and females must be using reliable contraception during the study and additionally for participants treated with ribavirin, for 6 months (for woman) and 7 months (for man and his partner) after treatment completion

Exclusion Criteria:

* Liver disease unrelated to HCV infection
* Hemoglobin (Hgb) <12g/dL in women and <13g/dL in men; white blood cells (WBC) <3,000/uL; platelets (PLTs) <100,000/ul
* Women with ongoing pregnancy or who are breast feeding
* History of severe psychiatric disease, especially depression
* History of neurologic disease, especially epilepsy
* History or evidence of symptoms of severe cardiac, gastrointestinal and kidney disease
* Positive anti-Human Immunodeficiency Virus (HIV) antibodies
* Positive anti-nuclear antibodies (ANA) and/or Anti-Smooth Muscle Antibody (ASMA) (>1/80)
* Positive Hepatitis B surface antigen (HBsAg)
* History of having received any systemic anti-neoplastic or immunomodulatory treatment in the previous 6 months
* History or other evidence of severe illness or any other conditions which would make the participants, in the opinion of investigator, unsuitable for the study (active drug addict except those under methadone treatment, thalassemic, dyalized included)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2003-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Santantonio T, Fasano M, Sagnelli E, Tundo P, Babudieri S, Fabris P, Toti M, Di Perri G, Marino N, Pizzigallo E, Angarano G; Acute Hepatitis C Study Group. Acute hepatitis C: a 24-week course of pegylated interferon alpha-2b versus a 12-week course of pegylated interferon alpha-2b alone or with ribavirin. Hepatology. 2014 Jun;59(6):2101-9. doi: 10.1002/hep.26991. Epub 2014 Apr 29. PMID 24442928

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 130 participants were randomized to pegylated-interferon alpha-2b at the dose of 1.5 mcg/kg/week for 24 weeks (PEG-IFN 24), pegylated-interferon alpha-2b at the dose of 1.5 mcg/kg/week for 12 weeks (PEG-IFN 12), or pegylated-interferon alpha-2b at the dose of 1.5 mcg/kg/week + ribavirin at the dose of 10.6 mg/kg/day for 12 weeks (PEG-IFN + RVB 12).
Groups:
- PEG-IFN + RVB 12: Pegylated interferon alpha-2b 1.5 ug/kg/week in combination with ribavirin 10.6 mg/kg/day for 12 weeks
Period: Treatment
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12
Started | 44 | 43 | 43
Completed Final Treatment Visit | 44 (Included 6 that discontinued the treatment before completion,but performed the Final Treatment Visit) | 43 (Included 3 that discontinued the treatment before completion,but performed the Final Treatment Visit) | 43 (Included 1 that discontinued the treatment before completion,but performed the Final Treatment Visit)
Completed | 38 | 40 | 42
Not Completed | 6 | 3 | 1
Not completed — Serious Adverse Event | 1 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Poor Protocol Compliance | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Period: Follow-up
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12
Started | 37 | 38 | 39
Completed | 29 | 28 | 29
Not Completed | 8 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12 | Total
Number analyzed (Participants) | 44 | 43 | 43 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.55 (13.86) | 38.32 (13.95) | 38.52 (12.48) | 37.79 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 6 | 37
  Male | 29 | 27 | 37 | 93
Region of Enrollment [Number; unit: participants]
  Italy | 44 | 43 | 43 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Response (SR) at the End of the 6-month Follow-up Period
Description: SR was defined as serum Hepatitis C Virus (HCV RNA) level at the end of 6-month follow-up below 15 IU/mL.
Time Frame: Evaluated at the end of 6 months
Population: Intent-to-treat population (ITT): including all randomized participants who received at least one dose of study medication. Participants without measurements at the end of treatment or who discontinued the study for any reason before the end of the treatment were considered as non-responders.
Measure: Number; unit: participants
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12
Number analyzed (Participants) | 44 | 43 | 43
participants | 23 | 20 | 21

2. Secondary Outcome: Virologic Response at the End of Treatment Follow-up (ETR)
Description: ETR was achieved if serum HCV RNA level at the end of 12 or 24 weeks
  treatment (depending on treatment arm) was <15 IU/mL.
Time Frame: At the end of treatment (either 12 weeks or 24 weeks depending on randomization).
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12
Number analyzed (Participants) | 44 | 43 | 43
participants | 26 | 28 | 27

3. Secondary Outcome: Virologic Response at 12 Months Post-treatment Follow-up (Long-term Response, [LTR]).
Description: LTR was obtained if serum HCV RNA level at the end of 12-month follow-up was <15 IU/mL.
Time Frame: At 12 months post-treatment (treatment period either 12 weeks or 24 weeks depending on randomization).
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12
Number analyzed (Participants) | 44 | 43 | 43
participants | 20 | 19 | 19

4. Secondary Outcome: Number of Participants Presenting With Alanine Transferase (ALT) Level Normalization
Description: ALT normalization was used as a measure of biochemical response to treatment. ALT levels were assessed at each study visit by the local laboratory, and efficacy measurements at the end of treatment, at 6 and 12 months post treatment follow-up were reported.
Time Frame: Evaluated at end of treatment (either 12 weeks or 24 weeks, depending on randomization), at 6-month follow-up visit, or at 12-month follow-up visit.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12
Number analyzed (Participants) | 44 | 43 | 43
participants
  End of Treatment | 28 | 31 | 32
  6-month Follow-up Period | 31 | 27 | 28
  12-month Follow-up Period | 27 | 23 | 23

5. Secondary Outcome: Number of Participants With Rapid Virologic Response (RVR)
Description: Participants were considered to have RVR if serum HCV RNA level at 2 or 4
  weeks of treatment was below the cut off value of the referring local
  laboratory of each participating site.
Time Frame: Evaluated at 2 and 4 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12
Number analyzed (Participants) | 44 | 43 | 43
participants
  2 weeks after start of treatment | 24 | 25 | 23
  4 weeks after start of treatment | 28 | 35 | 34

6. Secondary Outcome: Number of Peripheral Blood Mononuclear Cells (PBMCs)
Description: Cellular Differentiation Cluster Antigen 8-Positive (CD8+) PBMCs were measured at randomization, Treatment Weeks 2, 4, 8, and 12.
Time Frame: Treatment Weeks 2, 4, 8, and 12
Population: The association between HCV specific immune and SR to be assessed applying descriptive methods could not be evaluated as PBMC measurements were not carried out.
Arm/Group | PEG-IFN 24 | PEG-IFN 12 | PEG-IFN + RVB 12
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | PEG-IFN 12 | PEG-IFN 24 | PEG-IFN + RVB 12
Serious Adverse Events (participants affected / at risk) | 3/43 | 4/44 | 4/43
Other Adverse Events (participants affected / at risk) | 37/43 | 43/44 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN 12 (N=43) | PEG-IFN 24 (N=44) | PEG-IFN + RVB 12 (N=43)
HypoAcusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Optic Neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pyschotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN 12 (N=43) | PEG-IFN 24 (N=44) | PEG-IFN + RVB 12 (N=43)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4)
Granulocytopenia (Blood and lymphatic system disorders) | 22 (25) | 32 (44) | 26 (34)
Leukopenia (Blood and lymphatic system disorders) | 31 (36) | 30 (45) | 31 (37)
Neutropenia (Blood and lymphatic system disorders) | 6 (7) | 3 (3) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (9) | 3 (4)
Asthenia (General disorders) | 12 (12) | 11 (11) | 7 (7)
Chills (General disorders) | 4 (4) | 1 (1) | 6 (6)
Irritability (General disorders) | 2 (2) | 4 (4) | 2 (2)
Pain (General disorders) | 8 (8) | 9 (9) | 7 (8)
Pyrexia (General disorders) | 27 (31) | 30 (35) | 28 (34)
Hemoglobin Decreased (Investigations) | 1 (1) | 7 (7) | 5 (5)
Platelet Count Decreased (Investigations) | 7 (7) | 5 (6) | 1 (1)
Transaminases Increased (Investigations) | 4 (4) | 8 (9) | 2 (2)
Weight Decreased (Investigations) | 0 (0) | 4 (4) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (15) | 13 (14) | 13 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 11 (11) | 13 (15) | 12 (14)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 6 (6) | 5 (6)
Insomia (Psychiatric disorders) | 1 (1) | 5 (5) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7) | 2 (2)
Erythrema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publish or present any results of the study without the prior written permission of Schering-Plough The principal investigator further agrees to allow the Sponsor to review, 30 days prior to submission for publication or presentation, copies of abstracts or manuscripts for publication (including texts of oral presentations) which report any results of the study.